CLINICAL TRIAL: NCT01703104
Title: The Effect of Jobelyn ( Extract of Sorghum Bicolor) on the Haematological Parameters of Patients With Sickle Cell Anaemia Disease.
Brief Title: The Efficacy of Jobelyn (Sorghum Bicolor Extract)in the Treatment of Sickle Cell Anemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Lagos State University (Other)
Responsible Party: Principal Investigator, Dr. A. O. Dosunmu, CONSULTANT IN THE DEPARTMENT OF HAEMATOLOGY & BLOOD TRANSFUSION, LASUTH, Lagos State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: LASUTH/SCD02/2012
Record Dates: First submitted 2012-10-03; First posted 2012-10-10 (Estimated); Last update posted 2012-10-10 (Estimated); Status verified 2012-10

CONDITIONS: Sickle Cell Anemia
Keywords: Sorghum bicolor; sickle cell anaemia; haematological parameters
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Proguanil; Folic Acid

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Paludrine + Folic Acid (Active Comparator): This arm uses routine drugs, Paludrine + Folic Acid
  Interventions: Drug: Paludrine + Folic Acid
- Paludrine + Folic Acid + Jobelyn (Active Comparator): This group uses Paludrine + Folic Acid + Jobelyn
  Interventions: Dietary Supplement: Paludrine + Folic Acid + Jobelyn

INTERVENTIONS:
Drug: Paludrine + Folic Acid — This is the combination of routine drugs for treating sickle cell disease
  Other Names: Routine drugs
  Arms: Paludrine + Folic Acid
Dietary Supplement: Paludrine + Folic Acid + Jobelyn — Combination of routine drugs + Jobelyn
  Other Names: 1. Routine Drugs, i.e. Paludirine + Folic Acid; 2. Sorghum bicolor extract (Jobelyn)
  Arms: Paludrine + Folic Acid + Jobelyn

SUMMARY:
The primary objective is to determine if there is a significant increase in the haematocrit value of patients on Jobelyn and standard therapy compared to those on standard therapy alone.

DETAILED DESCRIPTION:
Sickle cell anaemia is an inherited haemoglobinopathy caused by a point missense mutation (GAG to GTG) in the beta globin gene that resulted in the substitution of an acidic amino acid ( glutamic acid) with a neutral and hydrophobic amino acid (valine) in the codon 6 of the beta globin chain. This genetic defect has a prevalence of 20% to 40% in Sub Saharan Africa, 7.8% in African Americans and to a lesser extent in the Middle East, Mediterranean and India.

The higher frequency in the sub Saharan Africa is thought to be due to the selective advantage the gene confers on the traits (heterozygotes state) in malaria zone. Nigeria is the most populous country in this region with about 24% frequency of the mutant gene. The prevalence of sickle cell anaemia in Nigeria is about 20 per 1000 life births. This implies that Nigeria may have the highest burden of the disease in the world.

The severity of sickle cell disease varies. The disease is more severe in patients with haemoglobin SS or haemoglobin S beta thalassaemia than in those with haemoglobin S beta+ thalassaemia or haemoglobin SC disease. The Arab - Indian haplotype produces a less severe disease than the African haplotype. Similarly, the coinheritance of one or two, alpha globin chain deletions or high fetal haemoglobin level in hereditary persistence of fetal haemoglobin are associated with mild disease, The severity is therefore higher in the Sub Saharan African sub region. However, the severity of the disease varies widely for unexplained reasons among patients with haemoglobin SS in this region.

The beta S globin chain binds at the valine site with complementary hydrophobic effects on other beta globin chain. This triggers the formation of polymers of haemoglobin. The rate of polymerization is increased with increase in intracellular deoxy-haemoglobin. Factors that promote polymerisation are dehydration, acidosis, increase in the level of 2,3 diphosphoglycerate which may occur in infections. On the other hand, the association of haemoglobin 5 with other haemoglobin that have higher oxygen affinity-like haemoglobin F or haemoglobin A reduce the rate of polymerisation.

The haemoglobin polymer forms a firm gel that damages the cellular membrane. The damaged membrane causes movement of potassium and water out of the cell thus leading to dehydration and more polymer formation. This damage also causes the negatively charged phosphatidylserine to move to the membrane surface and the red cell becomes deformed in shape, more rigid and more adherent to the vascular endothelium. The result of these are easy fragmentation of the membrane and extra vascular haemolysis, complement mediated lysis of the cell and intravascular haemolysis, shortened red cell survival to 4 to 25 days, trapping of rigid irreversible sickle cells in the post capillary venules which is promoted by leukocytosis, platelet activation and inflammatory cytokines.

The release of intravascular haemoglobin mobs up nitric acid which has a vasodilatation effect. This aggravates the already deficient tissue perfusion. A vicious circle is formed that eventually leads to tissue hypoxia, sequestration of blood in organs with sinuses (spleen, liver, lungs and the penis). There is also a chronic haemolytic anaemia with insufficient increase in the production of erythropoietin due to the fact that the beta S globin chain has a lower affinity for oxygen and therefore releases oxygen easily to the tissue. To further reduce erythropoiesis is the increase of inflammatory cytokines that inhibit haemopoiesis i.e interleukin 1 and tumor necrotic factor. On the other hand an increase in the red cell mass tends to increase vascular occlusion and ischemic crises. The ideal stable haematocrit for sickle cell disease is therefore between 24% and 28%. At this range of haematocrit, tissue hypoxia is minimized and painful crises are easier to control.

Factors that precipitate crises are dehydration, infection, extreme heat or cold and physical or emotional stress. These factors are prevalent in our environment. Early detection and preventive measures are very important in the management of sickle cell disease. To enhance red cell production, patients are offered regular folic acid. To prevent malaria, prophylactic paludrine is given and infection is treated with appropriate antibiotic. Among the anti sickling drugs, hydroxyurea, an inhibitor of ribonucleotide reductase, has been shown to decrease the rate of painful crises probably by reducing adhesion to the endothelium, increasing the proportion of fetal haemoglobin within the cell and reduction in the white blood cells and platelets. Other drugs on trial are butyrate compounds and analogues of azacytidine.

Other modalities are blood transfusion, exchange blood transfusion, stem cell transplant and the possibility of gene therapy is realistic. These modalities are not without their side effects and high costs. A new drug added to the routine drugs might minimize tissue. Hypoxia, rate of sickling and haemolysis if the haematocrit is within the steady state range, white cells count are reduced and inflammatory cytokines are reduced.

Available reports suggest that sickle cell erythrocytes are susceptible, to endogenous free radical mediated oxidative damage as indicated by marked increase in lipid peroxidation and superoxide dismutase level in haemoglobin SS patient. However there remain discrepancies in the status of anti oxidant enzymes and vitamins in the patients.

Sorghum bicolor, a grain long used in Africa for its high nutritional value also exhibits strong antioxidant properties and antiinflammatory effects. The traditional preparation of Sorghum bicolor has an oxygen radical absorbance capacity (ORAC) OF 3,123 micro mole TE/g. This is much higher than other botanical preparations. Complementing the antioxidant properties, sorghum bicolor also exhibits anti inflammatory effects and demonstrated selective COX-2 inhibition, providing effective reduction in inflammation without residual side effects.

Sorghum bicolor extract has been shown to increase the haematocrit and haemoglobin level and reduce the white cell count in trypanosome brucei brucei induced anaemia in experimental rabbits. These effects were conclusive within 49 days of experimentation. Animals sacrificed after the administration of lethal dose Jobelyn were shown to have congestion of the liver, kidneys and lungs. This might be as a result of direct effect on these organs or a sign of cardiotoxicity. However there is a wide therapeutic range.

Jobelyn is the proprietary name for the product intended to treat sickle cell disease and it is currently marketed as a nutritional supplement. Jobelyn is marketed in 250mg capsules of Sorghum bicolor leaf extract. The product is widely marketed in many countries including Nigeria. Many of our sickle cell patients have been using it regularly for a long time without any report of adverse effect.

The sorghum bicolor extract is expected to increase the haematocrit of' sickle cell anaemia within a short time, to reduce leukocytosis during sickling and therefore reduce vascular occlusion and improve tissue perfusion. The selective effect on COX 2 and the moderation of inflammatory cytokines is expected to reduce painful crises and inhibition of haemopoiesis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 14 to 45 years of age
* Haemoglobin SS

Exclusion Criteria:

* Patients with chronic inflammatory disease like tuberculosis
* Patients with chronic viral hepatitis or positive for human immunodeficiency virus
* Patients with autoimmune disorders.

  . patients with other haemoglobinopathy
* Pregnancy or anticipated pregnancy.
* Patient on drug abuse or alcohol abuse.
* Patients on treatment for organ failure

Ages: 14 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Actual)
Dates: Start 2012-01; Primary Completion 2012-03 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events | 12 weeks
  The number of participants who reported with Adverse events for the 12-week duration of the study

SECONDARY OUTCOMES:
number of blood transfusions during the 12-week trial period | 12 weeks
  No of blood transfusions carried out during the period as a result of anaemia

CONTACTS AND LOCATIONS:
Overall Officials: A O Dosunmu, M.D., Principal Investigator — Lagos State University
Locations (1):
- Lagos State University Teaching Hospital, Ikeja, Lagos, Nigeria

REFERENCES:
- [Background] Brohan M, Jerkovic V, Collin S. Potentiality of red sorghum for producing stilbenoid-enriched beers with high antioxidant activity. J Agric Food Chem. 2011 Apr 27;59(8):4088-94. doi: 10.1021/jf1047755. Epub 2011 Mar 7. PMID 21381750
- [Background] Geera B, Ojwang LO, Awika JM. New highly stable dimeric 3-deoxyanthocyanidin pigments from sorghum bicolor leaf sheath. J Food Sci. 2012 May;77(5):C566-72. doi: 10.1111/j.1750-3841.2012.02668.x. Epub 2012 Apr 10. PMID 22489620
- [Background] Kayode AP, Nout MJ, Linnemann AR, Hounhouigan JD, Berghofer E, Siebenhandl-Ehn S. Uncommonly high levels of 3-deoxyanthocyanidins and antioxidant capacity in the leaf sheaths of dye sorghum. J Agric Food Chem. 2011 Feb 23;59(4):1178-84. doi: 10.1021/jf103963t. Epub 2011 Jan 25. PMID 21322653
- [Background] Yang L, Browning JD, Awika JM. Sorghum 3-deoxyanthocyanins possess strong phase II enzyme inducer activity and cancer cell growth inhibition properties. J Agric Food Chem. 2009 Mar 11;57(5):1797-804. doi: 10.1021/jf8035066. PMID 19256554
- [Background] Shih CH, Siu SO, Ng R, Wong E, Chiu LC, Chu IK, Lo C. Quantitative analysis of anticancer 3-deoxyanthocyanidins in infected sorghum seedlings. J Agric Food Chem. 2007 Jan 24;55(2):254-9. doi: 10.1021/jf062516t. PMID 17227050
- [Background] Hunt DM, Emerson SU, Wagner RR. RNA- temperature-sensitive mutants of vesicular stomatitis virus: L-protein thermosensitivity accounts for transcriptase restriction of group I mutants. J Virol. 1976 May;18(2):596-603. doi: 10.1128/JVI.18.2.596-603.1976. PMID 178900
- [Background] Burdette A, Garner PL, Mayer EP, Hargrove JL, Hartle DK, Greenspan P. Anti-inflammatory activity of select sorghum (Sorghum bicolor) brans. J Med Food. 2010 Aug;13(4):879-87. doi: 10.1089/jmf.2009.0147. PMID 20673059
- [Background] Park JH, Darvin P, Lim EJ, Joung YH, Hong DY, Park EU, Park SH, Choi SK, Moon ES, Cho BW, Park KD, Lee HK, Kim MJ, Park DS, Chung IM, Yang YM. Hwanggeumchal sorghum induces cell cycle arrest, and suppresses tumor growth and metastasis through Jak2/STAT pathways in breast cancer xenografts. PLoS One. 2012;7(7):e40531. doi: 10.1371/journal.pone.0040531. Epub 2012 Jul 6. PMID 22792362
- [Background] Wu L, Huang Z, Qin P, Yao Y, Meng X, Zou J, Zhu K, Ren G. Chemical characterization of a procyanidin-rich extract from sorghum bran and its effect on oxidative stress and tumor inhibition in vivo. J Agric Food Chem. 2011 Aug 24;59(16):8609-15. doi: 10.1021/jf2015528. Epub 2011 Jul 29. PMID 21780844
- [Background] Awika JM, McDonough CM, Rooney LW. Decorticating sorghum to concentrate healthy phytochemicals. J Agric Food Chem. 2005 Aug 10;53(16):6230-4. doi: 10.1021/jf0510384. PMID 16076098
- [Background] Gee L, Abbott J, Conway SP, Etherington C, Webb AK. Validation of the SF-36 for the assessment of quality of life in adolescents and adults with cystic fibrosis. J Cyst Fibros. 2002 Sep;1(3):137-45. doi: 10.1016/s1569-1993(02)00079-6. PMID 15463820
- [Background] Okochi,V.I.,Okpuzor J, Okubena M.O., Awoyemi A.K. 2003 . The Influence of African Herbal Formula on the haematological parameters of trypanosome infected rats. African Journal of Biotechnology. 2 (9), 312-316.
- [Background] Erah P,O., Asonye C.C. Okhamafe A.O. 2003. Response of trypanosome brucei brucei induced anaemiato a commercialherbal preparation. African Journal of Biotechnology. 2,9, 307-311.
- [Background] Ogwumike OO. Hemopoietic effect of aqueous extract of the leaf sheath of Sorghum bicolor in albino rats. African Journal of Biomedical. Research. (2002): Vol 5; 69 - 71
- [Background] Oladiji AT, Jacob TO, Yakubu MT. Anti-anaemic potentials of aqueous extract of Sorghum bicolor (L.) moench stem bark in rats. J Ethnopharmacol. 2007 May 22;111(3):651-6. doi: 10.1016/j.jep.2007.01.013. Epub 2007 Jan 18. PMID 17306481
- [Background] Akande IS, Oseni AA, Biobaku OA. Effects of aqueous extract of Sorghum bicolor on hepatic, histological and haematological indices in rats. Journal of Cell and Animal Biology 4(9), 137-142, 2010.
- [Background] Nwinyi FC, Kwanashie HO. Evaluation of aqueous methanolic extract of Sorghum bicolor leaf base for antinociceptive and anti-inflammatory activities. African Journal of Biotechnology, 8 (18), 4642-4649, 2009.
- [Background] Eniojukan JF, Bolajoko AA. Toxicological Profiles of Commercial Herbal Preperation, Jobelyn. International Journal of Health Research, 2(4), 369-374, 2009.
- [Background] USDA Database for the Oxygen Radical Absorbance Capacity (ORAC) of Selected Foods, Release 2, U.S. Department of Agriculture, 2010.